CLINICAL TRIAL: NCT00394095
Title: A Double-Blind, Randomized, Placebo-Controlled, Pilot Study of Topiramate vs. Placebo in Combination With Olanzapine for the Prevention of Weight Gain in Manic or Mixed Youth With Bipolar Disorder
Brief Title: Topiramate vs. Placebo in Preventing Weight Gain in Bipolar Disorder Treated With Olanzapine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Melissa Delbello, Professor, University of Cincinnati
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: F1D-MC-X304
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Disorder; Weight Gain
Keywords: Bipolar Disorder; Weight Gain
MeSH Terms: conditions — Bipolar Disorder; Weight Gain | interventions — Topiramate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate Group (Experimental): Patients' initial dose of topiramate 25mg bid, which was titrated over 18 days to 150 mg bid (with flexibility to titrate to 200mg bid) as tolerated.
  Interventions: Drug: Topiramate
- Placebo Group (Placebo Comparator): Sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — Oral topiramate 300-400mg/day for 12 weeks
  Other Names: Topamax
  Arms: Topiramate Group
Drug: Placebo — Matched placebo to Experimental arm
  Other Names: Sugar pill
  Arms: Placebo Group

SUMMARY:
The primary objective of this study is to examine the efficacy of topiramate in combination with olanzapine for the prevention of weight gain in youth with bipolar disorder. The secondary objective is to examine the tolerability of topiramate in combination with olanzapine for the prevention of weight gain in youth with bipolar disorder.

DETAILED DESCRIPTION:
After consent and screening, patients will be initiated on 5mg or 10mg per day of olanzapine. Olanzapine doses will be titrated to 10-20 mg of olanzapine over one week, to a maximum of 20mg by day 21. Patients will also receive either topiramate (25mg bid titrated over 18 days to 150 mg bid. with flexibility to titrate to 200mg bid) or matched placebo. Topiramate will be initiated at a dose of 25 mg bid and will be increased by 25 mg bid every three days as tolerated. Patients will be evaluated by a blinded (to treatment status and adverse events) rater.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, ages 10-18 years.
2. Female patients of menarche must be using a medically accepted means of contraception (e.g. oral contraceptives, Depo-Provera, abstinence).
3. Each patient's authorized legal guardian must understand the nature of the study and must provide written informed consent. Each patient must also give assent to study participation.
4. Patients must have a diagnosis of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV-TR) bipolar disorder, type I and currently display an acute manic or mixed episode as determined by K-SADS (Geller et al 2000).
5. Patients must have a baseline (day 0) Young Mania Rating Scale score of at least 16.
6. Subjects should be fluent in English.

Exclusion Criteria:

1. Female patients who are either pregnant or lactating.
2. Clinically significant or unstable hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, hematologic or other systemic medical conditions.
3. Any history of current or past diabetes that has been treated with pharmacological intervention.
4. Neurological disorders including epilepsy, stroke, or severe head trauma.
5. Clinically significant laboratory abnormalities (> 3 times upper limit of normal), on any of the following tests: CBC with differential, electrolytes, BUN, creatinine, hepatic transaminases, lipid profile, fasting glucose, urinalysis, or thyroid indices. Clinically abnormal ECG.
6. Manic or mixed episode due to a general medical condition or substance-induced mania (DSM-IV-TR).
7. Mental retardation (IQ <70).
8. History of hypersensitivity to or intolerance of olanzapine or topiramate.
9. Prior history of olanzapine or topiramate non-response or allergic reaction.
10. DSM-IV substance (except nicotine or caffeine) dependence within the past 3 months.
11. Judged clinically to be at suicidal risk (defined as having active suicidal ideation, intent or plan, or a serious suicide attempt within 30 days, or a baseline Children's Depression Rating Scale suicide score of >3).
12. Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections and day 0.
13. Treatment with concurrent mood stabilizers or anticonvulsants, benzodiazepines (except as described below), psychostimulants, guanethidine, or guanadrel, or antidepressants.
14. Schizophrenia or other psychotic disorders (including schizophreniform disorder, schizoaffective disorder, delusional disorder, brief psychotic disorder, shared psychotic disorder, psychotic disorder due to a general medical condition, substance-induced psychotic disorder, psychotic disorder not otherwise specified) as defined in the DSM-IV.
15. Major depressive disorder, dysthymic disorder, depressive disorder not otherwise specified.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2006-12; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa P DelBello, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] DelBello MP, Bruns KM, Bloom T, Patino Duran LR, Strawn J, Adler CM, Welge J. A Double-Blind Placebo-Controlled Pilot Study of Topiramate in Manic Adolescents Treated with Olanzapine. J Child Adolesc Psychopharmacol. 2023 May;33(4):126-133. doi: 10.1089/cap.2022.0098. Epub 2023 May 2. PMID 37130314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty one bipolar adolescents with a manic or mixed episode (ages 12-18 years) were recruited from the inpatient units and outpatient clinics at the University of Cincinnati and Cincinnati Children's Hospital Medical Center.
Pre-assignment Details: Subjects meeting the entry criteria were randomized to treatment with topiramate or placebo in combination with olanzapine for this 12-week study.
Groups:
- Experimental Group: Topiramate Group: Experimental Group Receiving oral Topiramate, 300-400mg/day for 12 weeks
- Comparator Group: Placebo Group: Placebo Group Receiving oral placebo 300-400mg/day for 12 weeks
Period: Screening
Arm/Group | Experimental Group: Topiramate Group | Comparator Group: Placebo Group
Started | 17 | 14
Completed | 16 | 14
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Randomized
Arm/Group | Experimental Group: Topiramate Group | Comparator Group: Placebo Group
Started | 16 | 14
Completed | 8 | 10
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Overdose | 1 | 0
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group: Topiramate Group | Comparator Group: Placebo Group | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 14 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.9) | 14.0 (2.0) | 14.3 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index (BMI)
Description: For all participants, BMI was computed using Change in BMI [kg/m2 (weight/height2)] over 12 weeks from Baseline to Week 12.
Time Frame: 12 weeks
Population: The analysis was per protocol based on change in BMI over 12 weeks in the Experimental sample (N=16) compared to the Placebo group (N=14).
Measure: Mean (95% Confidence Interval); unit: kg/m2
Groups:
- Experimental Group: Topiramate Group: Change in Body Weight in kilograms over 12 weeks in the Experimental Topiramate sample (N=16) compared to the Placebo group (N=14).
- Placebo Group: Group receiving comparable dosage of placebo over 12 weeks.
Arm/Group | Experimental Group: Topiramate Group | Placebo Group
Number analyzed (Participants) | 16 | 14
kg/m2 | 0.8 [-.33 to 2.33] | 1.8 [1.20 to 11.72]

2. Primary Outcome: Change in Body Weight
Description: For all participants, change in body weight in kg over 12 weeks from Baseline to Week 12.
Time Frame: 12 weeks
Population: Bipolar youth (ages 12-17) who were taking olanzapine (10-20 mg/day) for a manic episode, were given topiramate (300-400mg/day) or comparable dose placebo for 12 weeks. Analysis was per protocol.
Measure: Mean (95% Confidence Interval); unit: kg
Groups:
- Comparator Group: Placebo Group: Group receiving comparable dosage of placebo over 12 weeks.
Arm/Group | Experimental Group: Topiramate Group | Comparator Group: Placebo Group
Number analyzed (Participants) | 16 | 14
kg | 2.8 [0.85 to 14.95] | 6.4 [0.85 to 14.95]

3. Secondary Outcome: Tolerability of Topiramate
Description: Maximum tolerated dosage of topiramate or placebo at end of study participation.
Time Frame: 12 weeks
Population: Bipolar youth (ages 12-17) who took at least one dose of study medication (topiramate or placebo).
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Experimental Group: Topiramate Group | Comparator Group: Placebo Group
Number analyzed (Participants) | 16 | 14
milligrams | 146.7 (67.4) | 175 (42.7)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events collected with open-ended questions and classified into categories by study team.
Arm/Group | Experimental Group: Topiramate Group | Comparator Group: Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/16 | 1/14
Other Adverse Events (participants affected / at risk) | 15/16 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group: Topiramate Group (N=16) | Comparator Group: Placebo Group (N=14)
Malignant hyperthermia (Nervous system disorders) | 1 (1) | 0 (0)
Increased aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group: Topiramate Group (N=16) | Comparator Group: Placebo Group (N=14)
Gastrointestinal (Gastrointestinal disorders) | 6 (6) | 5 (5)
Earache (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Muscle aches (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Upper extremity paresthesia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Headaches (General disorders) | 6 (6) | 5 (5)
Chest pain (General disorders) | 0 (0) | 3 (3)
Back and/or neck pain (General disorders) | 3 (3) | 1 (1)
Ocular/visual blurriness (Eye disorders) | 3 (3) | 1 (1)
Worsening of mood (Psychiatric disorders) | 2 (2) | 1 (1)
Sedation (Psychiatric disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes